CLINICAL TRIAL: NCT00429364
Title: Trial of Beta Blocker Therapy (Atenolol) Versus Angiotensin II Receptor Blocker Therapy (Losartan) in Individuals With Marfan Syndrome (A Trial Conducted by the Pediatric Heart Network)
Brief Title: Comparison of Two Medications Aimed at Slowing Aortic Root Enlargement in Individuals With Marfan Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); FDA Office of Orphan Products Development (U.S. Federal Agency); National Marfan Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 461; U01HL068270 (NIH)
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2014-01

CONDITIONS: Marfan Syndrome
Keywords: Aortic Root Dissection; Aortic Root Dilation; Pediatric Heart Network
MeSH Terms: conditions — Marfan Syndrome; Dissection, Ascending Aorta | interventions — Losartan; Atenolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atenolol (Active Comparator): Participants with Marfan's syndrome and ≥3 maximum aortic root z-score received 0.5 - 4.0 mg/kg/day Atenolol (not to exceed a total dose of 250 mg), with a goal of a 20% or greater decrease in the mean heart rate.
  Interventions: Drug: Atenolol
- Losartan (Active Comparator): Participants with Marfan's syndrome and ≥3 maximum aortic root z-score received 0.4 - 1.4 mg/kg/day Losartan (not to exceed a total dose of 100 mg).
  Interventions: Drug: Losartan Potassium

INTERVENTIONS:
Drug: Losartan Potassium — Losartan .3 - 1.4 mg/kg
  Other Names: Cozaar
  Arms: Losartan
Drug: Atenolol — Atenolol .5 - 4 mg/kg
  Other Names: Tenormin
  Arms: Atenolol

SUMMARY:
Marfan syndrome is a hereditary connective tissue disorder. Many individuals with this condition die because of the associated heart and blood vessel abnormalities. This study will compare the effectiveness of two medications, losartan and atenolol, at slowing aortic root enlargement in individuals with Marfan syndrome.

DETAILED DESCRIPTION:
Marfan syndrome is an inheritable disorder that affects the body's connective tissue. An abnormal protein results in connective tissue that is weaker than normal. Because connective tissue is found throughout the body, Marfan syndrome can affect many body systems, including the skeleton, eyes, nervous system, skin, lungs, heart, and blood vessels. Overall, heart and blood vessel abnormalities are the leading cause of death in individuals with Marfan syndrome. A common blood vessel abnormality associated with this disease involves the aorta, which is the large artery that carries blood away from the heart to the rest of the body. The aortic root, the portion of the aorta that is attached to the heart, may enlarge and tear or even rupture. A tear or rupture is considered a life-threatening emergency. Recent studies have shown that the medication losartan may reduce aortic root growth and improve heart function. The purpose of this study is to compare the effectiveness of losartan versus atenolol at slowing aortic root growth in individuals with Marfan syndrome.

This 3-year study will enroll individuals with Marfan syndrome. Participants will be randomly assigned to receive either losartan or atenolol on a daily basis. All participants will initially receive a low dose of their assigned medication. This dose will be gradually increased every 3 to 4 weeks until the maximum tolerated dose is reached. A continuous electrocardiogram (ECG) that monitors heart rate and activity in 24-hour intervals will be used to determine the proper dose increase for each participant. Participants will then receive the maximum tolerated dose for the remainder of the study. Study visits will occur at baseline and Months 6, 12, 24, and 36. Each study visit will include a physical examination, a medical history review, an ECG, an echocardiogram, and questionnaires. Additionally, at the baseline study visit blood will be collected for laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Marfan syndrome, according to Ghent criteria (more information can be found in Appendix D of the protocol)
* Aortic root Z-score greater than 3.0

Exclusion Criteria:

* Prior aortic surgery
* Aortic root dimension at the sinuses of Valsalva greater than 5 cm
* Planned aortic surgery within 6 months of study entry
* Aortic dissection
* Shprintzen-Goldberg syndrome
* Loeys-Dietz syndrome
* Therapeutic (i.e., for arrhythmia, ventricular dysfunction, or valve regurgitation) rather than prophylactic use of angiotensin-converting enzyme (ACE) inhibitor, beta-blocker, or calcium channel blocker
* History of angioedema while taking an ACE inhibitor or beta-blocker
* Intolerance to losartan or other angiotensin II receptor blocker (ARB) that resulted in termination of therapy
* Intolerance to atenolol or other beta-blocker that resulted in termination of therapy
* Kidney dysfunction (i.e., creatinine greater than the upper limit of age-related normal values)
* Asthma of sufficient severity to prohibit the use of a beta-blocker
* Chronic use of steroids and/or beta-adrenergic agents with exacerbations of asthma that are frequent (averaging three or more per year) or severe (requiring hospitalization)
* Diabetes mellitus
* Pregnant or planning to become pregnant within 36 months of study entry
* Inability to complete study procedures, including history of poor acoustic windows (i.e., inability to obtain accurate measurement of aortic root)

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 608 (Actual)
Dates: Start 2007-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Lacro, MD, Principal Investigator — Boston Children's Hospital
Locations (26):
- United States (24):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Rady Children's Hospital / UCSD, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Minnesota - St. Paul, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia College of Physicians and Surgeons, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Ghent University Hospital, Ghent, Gent, Belgium
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hoskoppal A, Menon S, Trachtenberg F, Burns KM, De Backer J, Gelb BD, Gleason M, James J, Lai WW, Liou A, Mahony L, Olson AK, Pyeritz RE, Sharkey AM, Stylianou M, Wechsler SB, Young L, Levine JC, Tierney ESS, Lacro RV, Bradley TJ; Pediatric Heart Network Investigators. Predictors of Rapid Aortic Root Dilation and Referral for Aortic Surgery in Marfan Syndrome. Pediatr Cardiol. 2018 Oct;39(7):1453-1461. doi: 10.1007/s00246-018-1916-6. Epub 2018 Jun 11. PMID 29948025
- [Derived] Lacro RV, Dietz HC, Sleeper LA, Yetman AT, Bradley TJ, Colan SD, Pearson GD, Selamet Tierney ES, Levine JC, Atz AM, Benson DW, Braverman AC, Chen S, De Backer J, Gelb BD, Grossfeld PD, Klein GL, Lai WW, Liou A, Loeys BL, Markham LW, Olson AK, Paridon SM, Pemberton VL, Pierpont ME, Pyeritz RE, Radojewski E, Roman MJ, Sharkey AM, Stylianou MP, Wechsler SB, Young LT, Mahony L; Pediatric Heart Network Investigators. Atenolol versus losartan in children and young adults with Marfan's syndrome. N Engl J Med. 2014 Nov 27;371(22):2061-71. doi: 10.1056/NEJMoa1404731. Epub 2014 Nov 18. PMID 25405392
- [Derived] Lacro RV, Guey LT, Dietz HC, Pearson GD, Yetman AT, Gelb BD, Loeys BL, Benson DW, Bradley TJ, De Backer J, Forbus GA, Klein GL, Lai WW, Levine JC, Lewin MB, Markham LW, Paridon SM, Pierpont ME, Radojewski E, Selamet Tierney ES, Sharkey AM, Wechsler SB, Mahony L; Pediatric Heart Network Investigators. Characteristics of children and young adults with Marfan syndrome and aortic root dilation in a randomized trial comparing atenolol and losartan therapy. Am Heart J. 2013 May;165(5):828-835.e3. doi: 10.1016/j.ahj.2013.02.019. Epub 2013 Mar 26. PMID 23622922
- See also: Click here for the Pediatric Heart Network Web site — http://www.pediatricheartnetwork.org
- See also: Click here for the National Marfan Foundation Web site — http://www.marfan.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2007 through February 2011, a total of 21 clinical centers enrolled 608 participants into the study.
Pre-assignment Details: For subjects on prophylactic therapy with atenolol or other BB, ARB, ACEi, or calcium-channel blocker, before the study, the drug will be weaned over a 14-day period. After that, a drug washout period of 14-21 days will take place before baseline assessment and randomization.
Period: Overall Study
Arm/Group | Atenolol | Losartan
Started | 303 | 305
Completed | 271 | 272
Not Completed | 32 | 33
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Physician Decision | 4 | 2
Not completed — Lost to Follow-up | 7 | 6
Not completed — Death | 0 | 1
Not completed — Underwent aortic root surgery | 10 | 18
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atenolol | Losartan | Total
Number analyzed (Participants) | 303 | 305 | 608
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (6.5) | 11.0 (6.2) | 11.2 (6.3)
Age, Customized [Number; unit: participants] — Young adults were defined as male participants who were 16 to 25 years of age and female participants who were 15 to 25 years of age.
  participants
    Young adult | 76 | 75 | 151
    Child | 227 | 230 | 457
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 119 | 242
  Male | 180 | 186 | 366
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data on race and ethnicity provided by the participant or a family member at the time of enrollment.
  Participants
    Hispanic or Latino | 36 | 46 | 82
    Not Hispanic or Latino | 266 | 259 | 525
    Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants] — Data on race and ethnicity provided by the participant or a family member at the time of enrollment.
  participants
    White | 266 | 260 | 526
    Black | 21 | 25 | 46
    Asian | 6 | 10 | 16
    Other | 10 | 10 | 20
Presence of causal FBN1 mutation [Number; unit: participants]
  Yes | 93 | 88 | 181
  No | 9 | 15 | 24
  Unknown | 201 | 202 | 403
Family history of Marfan [Number; unit: participants]
  Yes | 180 | 181 | 361
  No | 115 | 109 | 224
  Unknown | 8 | 15 | 23
Maximum aortic-root diameter, cm [Mean (Standard Deviation); unit: centimeter] — Data are based on readings at a central echocardiographic laboratory. Echocardiographic data were missing for one participant in the losartan group because of an unreadable echocardiogram.
  centimeter | 3.4 (0.7) | 3.4 (0.7) | 3.4 (0.7)
Maximum aortic-root diameter z-score [Median (Inter-Quartile Range); unit: z-score] — Data are based on readings at a central echocardiographic laboratory. Echocardiographic data were missing for one participant in the losartan group because of an unreadable echocardiogram.
  z-score | 4.0 [3.5 to 4.8] | 4.0 [3.3 to 5.0] | 4.0 [3.4 to 4.9]
Maximum aortic-root diameter z-score [Number; unit: participants] — Data are based on readings at a central echocardiographic laboratory. Echocardiographic data were missing for one participant in the losartan group because of an unreadable echocardiogram.
  participants
    ≥z-score of 4.5 | 106 | 114 | 220
    <z-score of 4.5 | 197 | 191 | 388
Had medical history of cardiac surgery [Number; unit: participants]
  Yes | 6 | 6 | 12
  No | 297 | 299 | 596
Had medical history of cardiovascular disorder [Number; unit: participants] — Cardiovascular disorder was defined by exercise intolerance, syncope; arrhythmia, hypertension, or hypotension requiring therapy; chest pain, shortness of breath; or other cardiovascular conditions.
  participants
    Yes | 39 | 36 | 75
    No | 264 | 269 | 533
Prior use of beta-blocker [Number; unit: participants]
  Yes | 173 | 171 | 344
  No | 130 | 134 | 264
Had medical history of endocrine disorder [Number; unit: participants] — Endocrine disorder was defined by either the use of hormone therapy to limit growth, delayed puberty.
  participants
    Yes | 7 | 0 | 7
    No | 296 | 305 | 601
Had medical history of neurodevelopmental disorder [Number; unit: participants] — Neurodevelopmental disorder was defined as attention deficit-hyperactivity disorder requiring therapy, developmental delay requiring therapy, learning disability requiring services, or other neurodevelopmental conditions.
  participants
    Yes | 56 | 61 | 117
    No | 247 | 244 | 491
Had medical history of psychiatric disorder [Number; unit: participants] — Psychiatric disorder was defined as depression requiring therapy, anxiety, or other psychiatric conditions.
  participants
    Yes | 23 | 16 | 39
    No | 280 | 289 | 569

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Change in Aortic Root (Sinuses of Valsalva) Body-surface-area-adjusted Z-score
Description: The rate of aortic root enlargement, expressed as the annual change in the maximum aortic-root-diameter z score indexed to body-surface area over a 3-year period following randomization
Time Frame: Up to 3 years following randomization.
Measure: Least Squares Mean (Standard Error); unit: z-score/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
z-score/year | -0.139 (0.013) | -0.107 (0.013)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis — P values are based on a linear regression mixed-effect model comparing slopes under compound symmetry, with adjustment for baseline

2. Secondary Outcome: Annual Rate of Change in Aortic Root (Sinuses of Valsalva) Absolute Dimension
Description: The rate of change in the absolute dimension of the aortic root over a 3-year period following randomization
Time Frame: Up to 3 years following randomization.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
cm/year | 0.069 (0.004) | 0.075 (0.004)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Annual Rate of Change in Ascending-aorta-diameter Z Score, Adjusted by Body-surface-area.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose ascending-aorta-diameter z scores were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: z-score/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 296 | 303
z-score/year | -0.140 (0.013) | -0.114 (0.013)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.15, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Annual Rate of Change in the Absolute Diameter of the Ascending Aorta
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose absolute dimensions of the ascending aorta were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 296 | 303
cm/year | 0.039 (0.004) | 0.044 (0.004)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Annual Rate of Change in Aortic-annulus-diameter Z Score, Adjusted by Body-surface Area
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose aortic-annulus-diameter z scores were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: z-score/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 302 | 304
z-score/year | -0.279 (0.018) | -0.175 (0.018)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Annual Rate of Change in the Absolute Diameter of the Aortic Annulus
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose absolute dimensions of the aortic annulus were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 302 | 304
cm/year | 0.015 (0.003) | 0.030 (0.003)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Annual Rate of Change in Total Aortic Proximal Regurgitant Jet Area Indexed to Body-surface-area
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose total aortic proximal regurgitant jet area indexes were measured at baseline or at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: (mm^2/m^2)/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 301 | 303
(mm^2/m^2)/year | 0.005 (0.003) | 0.001 (0.003)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Annual Rate of Change in Weight
Time Frame: Up to 3 years following randomization.
Measure: Least Squares Mean (Standard Error); unit: kg/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
kg/year | 0.239 (0.153) | 0.229 (0.154)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.96, Mixed Models Analysis — Regression model adjusted for age at study visit

9. Secondary Outcome: Annual Rate of Change in Weight-for-age Z-score
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who were between 0-20 years of age and whose weight-for-age z-scores were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: z-score/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 270 | 278
z-score/year | 0.011 (0.013) | 0.019 (0.013)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.45, Mixed Models Analysis

10. Secondary Outcome: Annual Rate of Change in Weight-for-height Z-score
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who were <120 cm in heights and whose weight-for-height z-scores were measured at baseline or at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: z-score/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 58 | 61
z-score/year | -0.001 (0.072) | -0.157 (0.076)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis

11. Secondary Outcome: Annual Rate of Change in Height
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose heights were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
cm/year | 0.822 (0.204) | 0.935 (0.202)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.65, Mixed Models Analysis

12. Secondary Outcome: Annual Rate of Change in Height-for-age Z-score
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who were between 0-20 years of age and whose heights were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: z-score/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 269 | 272
z-score/year | 0.046 (0.013) | 0.019 (0.013)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis

13. Secondary Outcome: Annual Rate of Change in Body Mass Index
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose body mass indexes were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2 per year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 283 | 295
kg/m^2 per year | 0.063 (0.044) | 0.076 (0.044)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis

14. Secondary Outcome: Annual Rate of Change in Body Mass Index for Age Z-score
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who were between 0-20 years of age and whose body mass index for age z-scores were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: z-score/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 250 | 263
z-score/year | 0.007 (0.022) | 0.021 (0.022)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.64, Mixed Models Analysis

15. Secondary Outcome: Annual Rate of Change in Arm Span to Height Ratio
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose arm span to height ratios were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: 1/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 301 | 303
1/year | 0.001 (0.001) | 0.001 (0.001)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.49, Mixed Models Analysis

16. Secondary Outcome: Annual Rate of Change in Upper to Lower Segment Ratio
Time Frame: Up to 3 years following randomization.
Population: All randomized participants whose upper to lower segment ratios were measured at baseline and at any of the follow-up visits.
Measure: Least Squares Mean (Standard Error); unit: 1/year
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 301 | 301
1/year | -0.014 (0.002) | -0.015 (0.002)
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.59, Mixed Models Analysis

17. Secondary Outcome: Number of Participants With Aortic Dissection.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number; unit: participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
participants | 0 | 2

18. Secondary Outcome: Event Rate of Aortic Dissection.
Description: Percentage of participants who had aortic dissection over a 3-year period following randomization.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
Percentage of participants | 0 [0 to 0] | 0.7 [0.2 to 2.7]
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.16, Log Rank

19. Secondary Outcome: Number of Participants With Aortic-root Surgery.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number; unit: participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
participants | 10 | 18

20. Secondary Outcome: Event Rate of Aortic-Root Surgery
Description: Percentage of participants who had aortic-root surgery over a 3-year period following randomization.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
Percentage of participants | 3.4 [1.9 to 6.3] | 6.0 [3.8 to 9.4]
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.13, Log Rank

21. Secondary Outcome: Number of Death.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number; unit: participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
participants | 0 | 1

22. Secondary Outcome: Event Rate of Death
Description: Percentage of participants who died over a 3-year period following randomization.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
Percentage of participants | 0 [0 to 0] | 0.3 [0 to 2.4]
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.32, Log Rank

23. Secondary Outcome: Number of Participants With the Composite Adverse Clinical Outcomes, Including Aortic Dissection, Aortic-root Surgery and Death.
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number; unit: participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
participants | 10 | 19

24. Secondary Outcome: Event Rate of the Composite Adverse Clinical Outcomes, Including Aortic Dissection, Aortic-root Surgery and Death.
Description: Percentage of participants who had aortic dissection, aortic-root surgery or death over a 3-year period following randomization
Time Frame: Up to 3 years following randomization.
Population: All randomized participants who received the treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
Percentage of participants | 3.4 [1.9 to 6.3] | 6.4 [4.1 to 9.8]
Statistical Analysis 1: Comparison: Atenolol vs Losartan; Test type: Superiority or Other; p = 0.10, Log Rank

25. Secondary Outcome: Adverse Drug Reactions Reported at the Baseline Visit
Time Frame: At baseline
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 303 | 305
participants
  Headache, any severity | 112 | 114
  Headache, bothersome | 10 | 10
  Fatigue, any severity | 84 | 105
  Fatigue, bothersome | 0 | 0
  Mood alterations, any severity | 54 | 49
  Mood alterations, bothersome | 7 | 3
  Behavior changes, any severity | 21 | 23
  Behavior changes, bothersome | 2 | 1
  Insomnia, any severity | 60 | 61
  Insomnia, bothersome | 2 | 2
  Nightmares, any severity | 52 | 53
  Nightmares, bothersome | 2 | 3
  Dizziness with standing, any severity | 60 | 58
  Dizziness with standing, bothersome | 0 | 2
  Dizziness - other, any severity | 25 | 27
  Dizziness - other, bothersome | 0 | 1
  Fainting with loss of consciousness, any severity | 5 | 9
  Fainting with loss of consciousness, bothersome | 5 | 9
  Palpitations, any severity | 60 | 53
  Palpitations, bothersome | 0 | 0
  Chest pain, any severity | 54 | 58
  Chest pain, bothersome | 1 | 5
  Dyspnea, any severity | 43 | 38
  Dyspnea, bothersome | 3 | 0
  Wheezing, any severity | 15 | 14
  Wheezing, bothersome | 2 | 1
  Upper respiratory/Nasal congestion, any severity | 106 | 117
  Upper respiratory/Nasal congestion, bothersome | 0 | 2
  Cough, any severity | 47 | 59
  Cough, bothersome | 1 | 0
  Dysgeusia, any severity | 10 | 3
  Dysgeusia, bothersome | 0 | 0
  Stomach pain/Indigestion, any severity | 47 | 61
  Stomach pain/Indigestion, bothersome | 0 | 1
  Nausea, any severity | 30 | 35
  Nausea, bothersome | 1 | 0
  Vomiting, any severity | 23 | 23
  Vomiting, bothersome | 0 | 0
  Diarrhea, any severity | 35 | 43
  Diarrhea, bothersome | 1 | 1
  Constipation, any severity | 44 | 35
  Constipation, bothersome | 0 | 0
  Vascular (hands, feet), any severity | 35 | 34
  Vascular (hands, feet), bothersome | 0 | 1
  Muscle pain or Cramps, any severity | 59 | 58
  Muscle pain or Cramps, bothersome | 2 | 4
  Back pain, any severity | 60 | 67
  Back pain, bothersome | 3 | 2
  Periorbital edema, any severity | 13 | 15
  Periorbital edema, bothersome | 0 | 0
  Pedal edema, any severity | 2 | 3
  Pedal edema, bothersome | 0 | 0
  Other, any severity | 21 | 16
  Other, bothersome | 3 | 1

26. Secondary Outcome: Adverse Drug Reactions Reported During Routine Follow-up Surveillance
Time Frame: From 6 months to 3 years following randomization.
Population: All subjects who had any of the follow-up visits after 6 months post-randomization.
Measure: Number; unit: participants
Arm/Group | Atenolol | Losartan
Number analyzed (Participants) | 291 | 297
participants
  Headache, any severity | 202 | 208
  Headache, bothersome | 27 | 20
  Fatigue, any severity | 152 | 153
  Fatigue, bothersome | 7 | 5
  Mood alterations, any severity | 89 | 86
  Mood alterations, bothersome | 13 | 13
  Behavior changes, any severity | 51 | 46
  Behavior changes, bothersome | 5 | 8
  Insomnia, any severity | 108 | 107
  Insomnia, bothersome | 6 | 4
  Nightmares, any severity | 100 | 94
  Nightmares, bothersome | 7 | 4
  Dizziness with standing, any severity | 119 | 105
  Dizziness with standing, bothersome | 6 | 0
  Dizziness - other, any severity | 60 | 61
  Dizziness - other, bothersome | 2 | 0
  Fainting with loss of consciousness, any severity | 21 | 16
  Fainting with loss of consciousness, bothersome | 21 | 16
  Palpitations, any severity | 86 | 101
  Palpitations, bothersome | 0 | 0
  Chest pain, any severity | 114 | 106
  Chest pain, bothersome | 14 | 1
  Dyspnea, any severity | 75 | 72
  Dyspnea, bothersome | 1 | 3
  Wheezing, any severity | 36 | 32
  Wheezing, bothersome | 2 | 5
  Upper respiratory/Nasal congestion, any severity | 188 | 186
  Upper respiratory/Nasal congestion, bothersome | 3 | 3
  Cough, any severity | 117 | 113
  Cough, bothersome | 1 | 1
  Dysgeusia, any severity | 29 | 16
  Dysgeusia, bothersome | 0 | 0
  Stomach pain/Indigestion, any severity | 119 | 121
  Stomach pain/Indigestion, bothersome | 2 | 8
  Nausea, any severity | 99 | 78
  Nausea, bothersome | 0 | 0
  Vomiting, any severity | 81 | 75
  Vomiting, bothersome | 1 | 2
  Diarrhea, any severity | 94 | 90
  Diarrhea, bothersome | 1 | 3
  Constipation, any severity | 77 | 66
  Constipation, bothersome | 1 | 0
  Vascular (hands, feet), any severity | 73 | 66
  Vascular (hands, feet), bothersome | 0 | 0
  Muscle pain or Cramps, any severity | 148 | 124
  Muscle pain or Cramps, bothersome | 6 | 7
  Back pain, any severity | 137 | 134
  Back pain, bothersome | 5 | 8
  Periorbital edema, any severity | 22 | 27
  Periorbital edema, bothersome | 0 | 1
  Pedal edema, any severity | 6 | 5
  Pedal edema, bothersome | 0 | 0
  Other, any severity | 105 | 108
  Other, bothersome | 10 | 12

ADVERSE EVENTS:
Time Frame: The adverse event (AE) data were collected since randomization till the end of the study, for up to 3 years.
Description: Serious AEs and important medical events (including pregnancy) were reported within 24 hours of first knowledge of event; Non-Serious AEs were reported within 7 calendar days of first knowledge of event.
Arm/Group | Atenolol | Losartan
Serious Adverse Events (participants affected / at risk) | 27/303 | 33/305
Other Adverse Events (participants affected / at risk) | 135/303 | 121/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atenolol (N=303) | Losartan (N=305)
Blood/bone marrow(sickle cell crisis) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (4)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis NOS (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Valvular heart disease NOS (Cardiac disorders) | 0 (0) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Autoimmune disorder NOS (Immune system disorders) | 1 (2) | 1 (1)
Hypersensitivity NOS (Immune system disorders) | 0 (0) | 1 (1)
Serum sickness (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 1 (1)
Respiratory tract infection NOS (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection NOS (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound - snake bite (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (2)
Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular: vessel injury-artery, other NOS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral abscess (Nervous system disorders) | 1 (2) | 0 (0)
Convulsions NOS (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Psychosis aggravated (Psychiatric disorders) | 1 (1) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7)
Pulmonary/upper respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Culture wound negative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic root enlargement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac General-other: mitral valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atenolol (N=303) | Losartan (N=305)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemoglobin (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac General - Other - Murmur (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac General - other - nonresponsive and pale (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 9 (9) | 10 (10)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Auditory/ear-other (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypersensitivity to sound (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hot flushes NOS (Endocrine disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 3 (3) | 1 (1)
Eyelid function disorder NOS (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Ocular-other (L eye burning/redness 4 mos. s/p lensectomy with lens insertion) (Eye disorders) | 1 (1) | 0 (0)
Ocular-other (right eye hemorrhage) (Eye disorders) | 1 (1) | 0 (0)
Ocular/Visual - Squinting of OS to see things more clearly. (Eye disorders) | 1 (1) | 0 (0)
Ocular/visual-other (redness and itching of eyes) (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain NOS (Gastrointestinal disorders) | 7 (7) | 7 (7)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diarrhoea NOS (Gastrointestinal disorders) | 4 (6) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal - HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oseophagitis NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peridontal disorder NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 5 (5) | 3 (3)
Tooth disorder NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting NOS (Gastrointestinal disorders) | 2 (3) | 5 (7)
Bilateral pedal edema (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 16 (18) | 17 (18)
Constitutional symptoms -other(flu) (General disorders) | 1 (1) | 0 (0)
Constitutional symptoms-other (unusual dreams) (General disorders) | 1 (1) | 0 (0)
Constitutional-other (general body cold sensation) (General disorders) | 0 (0) | 1 (1)
Edema:head and neck (General disorders) | 2 (2) | 2 (2)
Edema:limb (General disorders) | 1 (1) | 1 (2)
Falling asleep (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 18 (19) | 11 (12)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Influenza-like illness (General disorders) | 1 (1) | 0 (0)
Nightmare (General disorders) | 7 (8) | 13 (13)
Pain-other (right hip pain) (General disorders) | 1 (1) | 0 (0)
Pain-other:chest pain/costochondritis (diagnosed in ER as costochondritis) (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (6) | 2 (2)
Allergy/Immunology - Other (rash) (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity NOS (Immune system disorders) | 0 (0) | 3 (3)
Abcessed tooth (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis NOS (Infections and infestations) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Infection - Eye NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other - Parvovirus (Infections and infestations) | 0 (0) | 1 (1)
Infection Pharnyx (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC-eye, NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC-middle ear (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC-pharynx (Infections and infestations) | 0 (0) | 2 (2)
Infection with unknown ANC-sinus (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC-upper ariway NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection-bladder(urinary) (Infections and infestations) | 0 (0) | 1 (1)
Infection-other (sinus, bronchitis, pharyngeal) (Infections and infestations) | 1 (1) | 0 (0)
Infection-other (skin on foot) (Infections and infestations) | 0 (0) | 1 (1)
Infection-other-Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Infection: Dental - Tooth (Infections and infestations) | 1 (1) | 0 (0)
Middle ear infection (Infections and infestations) | 1 (1) | 2 (2)
Mononucleosis (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Sinus infection (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis NOS (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Vaginitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection coxsackievirus (Infections and infestations) | 1 (1) | 0 (0)
Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Joint disorder NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Msk/soft tissue, other (Nodule on back) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal (other) (loose joints-causing pain) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal/soft tissue - other (patellar dislocation) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal/soft tissue-other (Bursa on left shoulder blade due to back brace) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal/soft tissue-other (nodule on back) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal/soft tissue-other( left arm pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Cognitive disorder (Nervous system disorders) | 2 (2) | 2 (2)
Convulsions NOS (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 29 (29) | 17 (18)
Dizziness upon standing (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 31 (36) | 18 (19)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia NOS (Nervous system disorders) | 0 (0) | 1 (1)
Neurology - other (Nervous system disorders) | 0 (0) | 2 (2)
Neurology-other (panic attacks) (Nervous system disorders) | 0 (0) | 1 (2)
Panick attack (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 13 (14) | 9 (9)
Syncope vasovagal (Nervous system disorders) | 2 (2) | 2 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Sexual/reproductive function-other (4.5 cm cyst on right ovary) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Sexual/reproductive function-other (abnormal pap smear) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 11 (12) | 3 (3)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 9 (11) | 2 (3)
Insomnia (Psychiatric disorders) | 10 (10) | 12 (12)
Mood alteration (Psychiatric disorders) | 1 (1) | 0 (0)
Neurology-other (expression of anger and sadness) (Psychiatric disorders) | 1 (1) | 0 (0)
Neurology-other (irritability) (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 6 (6) | 3 (3)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/genitourinary-increased urinary frequency, daytime only, associated w/ po water intake (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0)
Urogenital haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7)
Hemorrhage/Bleeding - other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Nasal conjestion/inf with unk ANC upper airway NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary/upper respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne NOS (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Burn on skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Derm/skin-other (Poison Ivy) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Derm/skin-other (mild chin rash) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Derm/skin-other (possible aczema) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Derm/skin-other (worsening of underlying hand skin disorder) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology - other - Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/skin-other (Poison Ivy) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/skin-other (cervical dysplasia) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/skin-other (papules on legs) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatology/skin-other (rash: nonspecific maculopapular rash) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash on torso and neck (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Sweating increased (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria NOS (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Cardiac general-chest tightness (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension NOS (Vascular disorders) | 1 (1) | 0 (0)
Hypotension NOS (Vascular disorders) | 0 (0) | 3 (3)
Raynaud's Phenomena (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The effect of losartan on TGF-β was not assessed. The study results do not apply to Marfan subjects whose BSA-adj. aortic-root z score is ≤3.

Subjects may find their treatment based on the appearance of the drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications and presentations resulting from studies from the PHN Network must be approved by the Publications and Presentations Committee before submission. The Sponsor (NERI) and funding agency (NHLBI) both are represented on the P&P Committee along with Network Investigators. Members of the P&P Committee can recommend changes to publications.